CLINICAL TRIAL: NCT01954849
Title: Assessment of Therapeutic Potential of a Novel Dental Probiotic in Pediatric Patients Affected by Gingivitis
Brief Title: Assessment of a Probiotic to Treat Gingivitis in Pediatric Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Integra Medical Inc. (Industry); University of Toronto (Other); University of Western Ontario, Canada (Other); Ontario Centres of Excellence (Industry)
Responsible Party: Principal Investigator, Peter Cadieux, Adjunct Professor, University of Western Ontario, Canada
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LG-001; 185428 (Other: Health Canada, Natural Health Products Directorate); OCE VIP #20964 (Other Grant/Funding Number: Ontario Centres of Excellence)
Record Dates: First submitted 2013-09-26; First posted 2013-10-07 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Gingivitis; Inflammation
Keywords: gingivitis; inflammation; plaque; orthodontics
MeSH Terms: conditions — Gingivitis; Inflammation; Plaque, Amyloid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic formulation (Experimental): Probiotic dissolving lozenge, at least 1 billion total CFU, taken at a certain prescribed regimen for 28 days.
  Interventions: Dietary Supplement: Probiotic formulation
- Placebo (Placebo Comparator): Placebo dissolving lozenge, with the exact same appearance as the treatment lozenge (including flavour, colour, shape and texture), and formulated with all the same ingredients except for the live bacteria, taken for 28 days at the same prescribed regimen as the probiotic lozenge.
  Interventions: Dietary Supplement: Probiotic formulation

INTERVENTIONS:
Dietary Supplement: Probiotic formulation

SUMMARY:
This study investigates the efficacy of a proprietary probiotic formulation comprising 6 strains of bacteria in reducing inflammation and gingivitis in pediatric patients between 11 and 18 years old undergoing orthodontics treatment. Patients will be recruited based on a prior diagnosis of mild to moderate gingivitis by gingival index score. Participants in this study will be randomly assigned to receive either the probiotic treatment or a placebo, both in the form of a dissolving lozenge; for which the placebo is exactly the same shape, texture, taste, and composition as the probiotic treatment, but does not contain the active probiotic ingredients. The lozenges are to be taken orally at a certain prescribed regimen for 28 days. Participants will be assessed for gingivitis scores, gum bleeding scores, plaque scores, overall periodontal health, and for precarious areas at baseline, 14, and 28 days. They will also be assessed for the same measures at day 56, following a 28-day wash-out phase. Plaque and saliva samples will be collected at all timepoints for in vitro analyses of changes in microbial pathogens and/or inflammatory cytokines.

ELIGIBILITY:
Inclusion criteria:

* Are male or female between the ages of 11 to 18 years
* Have mild to moderate gingivitis as determined by dentist (GI of at least 1 to a maximum of 2)
* Are undergoing fixed orthodontic therapy on both arches with attachments on at least 20 teeth including bonded 1st molars for a minimum of 5 months.
* Have fully erupted teeth #16, #21, #23, #36, #41, and #43
* Are caries inactive prior to study initiation.
* Are in a healthy systemic condition
* Have not used any antimicrobial mouth rinses, probiotics (unrelated to the study), antibiotics or anti-inflammatories medications with one month prior to and during the study
* Whose legal guardian has given informed consent to participate in the study and must be able to communicate in English

Exclusion Criteria:

* Unable to make informed consent
* Subjects with allergies to milk or milk products, gluten or soy or any other ingredients present in the lozenge
* Immune compromised
* Major underlining medical condition
* Pregnancy
* History of smoking or alcohol consumption
* Have major dental conditions such as periodontal disease, dental caries and/or xerostemia or systemic diseases which could directly or indirectly affect plaque formation
* Use of medications within 1 month (antibiotics, anti-inflammatory, mouth rinses) that can influence the outcome.
* Ongoing or recent (within 1 month) use of probiotics unrelated to the study
* Have within the past 30 days experienced any nausea, fever, vomiting, bloody diarrhea or severe abdominal pain

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2014-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Reduction in gingivitis | 0, 14, 28, and 56 days
  Gingivitis will be assessed by gingival index:
  0 - Absence of gingival inflammation
  1. - Mild inflammation: slight change in colour, little change in texture of any portion of but not the entire marginal or papillary gingival unit
  2. - Mild inflammation: criteria as above, but involving the entire marginal or papillary gingival unit
  3. - Moderate inflammation: glazing, redness, edema, and/or hypertrophy of the marginal or papillary gingival unit
  4. - Severe inflammation: marked redness, edema, and/or hypertrophy of marginal or papillary gingival unit; spontaneous bleeding, congestion or ulceration.

SECONDARY OUTCOMES:
Reduced plaque | 0, 14, 28, and 56 days
  Reduction in levels of plaque as measured by a plaque index:
  0 - No plaque in the gingival area
  1. - A film of plaque adhering to the free gingival margin and adjacent area of the tooth, which can not be seen with the naked eye. Only seen by running a probe across the tooth surface
  2. - Moderate accumulation of plaque deposits within the gingival pocket, on the gingival margin and/ or adjacent tooth surface, which can be seen with the naked eye
  3. - Abundance of soft matter within the gingival pocket and/or on the gingival margin and adjacent tooth surface
Reduction in inflammation | 0, 14, 28, and 56 days
  Reduction in salivary cytokines IL-1, IL-6, IL-8, TNF-A, IL-12 and an increase in IL-10, and IL-13 as measured by immunofluorometric assay.

OTHER OUTCOMES:
Reduction in S. mutans | 0, 14, 28, and 56 days
  Reduced levels of S. mutans in plaque and saliva

CONTACTS AND LOCATIONS:
Overall Officials: Peter Cadieux, PhD, Principal Investigator — University of Western Ontario, Canada; Siew-Ging Gong, BDS, MS, MA, PhD., Study Director — University of Toronto, Canada
Locations (1):
- University of Toronto Orthodontics Clinic, Toronto, Ontario, Canada